CLINICAL TRIAL: NCT04630197
Title: Using Electronically Delivered Cognitive Behavioural Therapy and Functional Magnetic Resonance Imaging to Understand the Pathophysiology of Obsessive-compulsive Disorder
Brief Title: Using Online Delivered Therapy and Brain Imaging to Better Understand OCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Callum Stephenson (Other)
Collaborators: Online PsychoTherapy Clinic (Other)
Responsible Party: Sponsor-Investigator, Callum Stephenson, Principle Investigator, MSc Candidate, Queen's University
Organization: Queen's University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 48144
Record Dates: First submitted 2020-11-05; First posted 2020-11-16 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Obsessive-Compulsive Disorder; Psychotherapy; MRI; fMRI; Cognitive Behavioural Therapy; Mental Health Care; Virtual; Online; Internet; Electronic
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- e-CBT (Experimental): 16 weekly sessions will be conducted through OPTT and consist of approximately 30 slides and interactive therapist videos. The content and format will mirror in-person CBT for OCD. The connection between thoughts, behaviours, emotions, physical reactions, and the environment will be a focus. Moreover, mindfulness, body scanning, self-care, goal setting, thinking errors, the 5-part model, thought records, and ERP will be incorporated. Slides will highlight different topics each week and include general information, an overview of skills, and homework on that topic. The homework will be submitted through OPTT and reviewed by therapists with personalized feedback provided within 3 days of submission. Weekly homework submission for feedback will be mandatory before being eligible for the next session. After each completion of the e-CBT program, participants will be interviewed to investigate their experience using OPTT and their perception of how the treatment went.
  Interventions: Behavioral: e-CBT

INTERVENTIONS:
Behavioral: e-CBT — The description is provided in the treatment arm description.

SUMMARY:
This study will implement an e-CBT program for OCD and observe its effects on brain activation levels using functional magnetic resonance imaging (fMRI). It is hypothesized that brain activation levels in the basal ganglia and frontal cortex will decrease following treatment. Individuals with OCD will be offered a 16-week e-CBT program with ERP mirroring in-person CBT content that will be administered through a secure online platform. Efficacy of treatment will be evaluated using clinically validated symptomology questionnaires at baseline, week 8, week 16, and at a 6-month follow-up. Using fMRI at baseline and post-treatment, brain activation levels will be assessed at resting state, and while exposed to anxiety-inducing images (i.e., dirty dishes if cleanliness is an obsession). The effects of treatment on brain activation levels and the correlation between symptom changes and activation levels will be analyzed.

DETAILED DESCRIPTION:
Study Design:

A non-randomized pilot study design will be employed. Functional magnetic resonance imaging (fMRI) will be conducted at baseline and post-treatment to evaluate activation level changes in the basal ganglia and frontal cortex. Clinically validated symptomology questionnaires will be used to evaluate treatment efficacy. Additionally, qualitative interviews will be conducted to gather personal demographic information as well as information regarding participant experience while using the online psychotherapy clinic. This study has been registered on the ClinicalTrials.Gov Protocol Registration and Results System (NCT04630197). Additionally, ethics approval has been obtained from the Queen's University Health Sciences and Affiliated Teaching Hospitals Research Ethics Board (HSREB).

Participants:

Participants (n = 10) will be recruited from family medicine and psychiatric clinics at Queen's University and Kingston Health Sciences Centre sites (Hotel Dieu Hospital and Kingston General Hospital) in Kingston, Ontario, Canada. Additionally, local and social media advertisements will be utilized. Participants will be enrolled in the study based on referrals from outpatient clinics, family doctors, as well as self-referrals. Those invited and interested in participating will have the study protocol explained along with an evaluation by a psychiatrist on the research team through a secured video appointment. Participants will be evaluated for a diagnosis of OCD based on the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) [48]. Once a diagnosis of OCD is confirmed and the participant is given written and verbal instructions on how to participate in the online therapy, informed consent will be obtained. Inclusion criteria include the following: between the ages of 18 and 65 years at the start of the study, a diagnosis of OCD according to DSM-5, competence to consent to participate, ability to speak and read English, and consistent and reliable access to the internet. Exclusion criteria include having any metal implants or additional factors deemed not safe to undergo an MRI scan, active psychosis, acute mania, severe alcohol or substance use disorder, and/or active suicidal or homicidal ideation. Additionally, if a participant is receiving another form of psychotherapy, they will be excluded from the study.

e-CBT Protocol: Weekly sessions of e-CBT will be conducted through the Online Psychotherapy Tool (OPTT), a secure, online, cloud-based mental health care delivery platform. These online sessions will consist of approximately 30 slides and interactive therapist videos, with 16 modules in total (1 module per week). The content and format of these online sessions will mirror in-person CBT for OCD. The connection between thoughts, behaviours, emotions, physical reactions, and the environment will be a focus. Moreover, mindfulness, body scanning, self-care, goal setting, thinking errors, the 5-part model, and thought records will be employed as techniques for participants. ERP will be incorporated into the e-CBT program as this is the first-line route of treatment. Slides will highlight different topics each week and include general information, an overview of skills, and homework on that topic. The homework included in each session will be submitted through OPTT and reviewed by therapists with personalized feedback provided within 3 days of submission. Weekly homework submission for feedback will be mandatory before being eligible for the next session. After each completion of the e-CBT program, participants will be interviewed to investigate their experience using OPTT and their perception of how the treatment went. Participants can access their therapy sessions from any device with internet access (desktop computer, laptop, cellphone, tablet) and can be run on a variety of internet browsers.

fMRI Protocol: All imaging procedures will occur at the Queen's University MRI Facility in Kingston, Ontario, Canada using a Siemens 3.0 Tesla whole-body MRI scanner with a standard coil. Scans will occur at baseline (pre-treatment), after week 16 (post-treatment, and at a 6-month follow-up. During scanning, participants will lay on the scanning table on their back, with their head resting on a foam pad to reduce movement. Appointments will be 1 hour.

Anatomical reference images will be captured initially. Following this, fMRI scans will occur while participants are shown neutral images and anxiety-inducing images (i.e., dirty dishes if cleanliness is an anxiety-inducing concept for a specific participant). The frontal cortex and basal ganglia will be the focuses of the imaging procedures as we are interested in the activation level changes during neural anxiety processing. These images will be standardized pictures from the International Affective Picture System (IAPS) that will be selected specifically for each patient by members of our research team.

Participants will be shown a total of 40 images (20 neutral, 20 anxiety-inducing; R = 0.5) during the fMRI scans. There will be 4 fMRI runs that occur in the following sequence:

* 5 neutral images (30s per image, 5s break between), 1-minute break, 5 anxiety-inducing images (30s per image, 5s break between), 1-minute break.
* 5 new anxiety-inducing images (30s per image, 5s break between), 1-minute break, 5 new neutral images (30s per image, 5s break between), 1-minute break.
* 5 new anxiety-inducing images (30s per image, 5s break between), 1-minute break, 5 new neutral images (30s per image, 5s break between), 1-minute break.
* 5 neutral images (30s per image, 5s break between), 1-minute break, 5 anxiety-inducing images (30s per image, 5s break between).

The images will be shown in sets (groups of 5) as opposed to intermingled as we hope this will produce a more sustained emotional state and allow for more distinct readings. The reasoning of the sets being repeated in the middle (back-to-back of the anxiety-inducing images in the example above) is for participants to not become as accustomed to the ordering. Moreover, we will change this ordering for every participant (i.e, The next participant would receive back-to-back sets of the neutral imaging in runs 2 and 3). This is done to counterbalance the imaging sets. Participants will be prompted to imagine themselves in the situations described in the images. The images will appear on a screen and then be reflected into the scanner for participants to view. 0.5% blood oxygen level-dependent (BOLD) signal difference between conditions (p < 10-6) will be considered a detectable change (eff = 0.005).

Anatomical reference images will be captured with the phase encoding direction collected sagitaly from anterior to posterior. These images will be captured with T1-weighted high-resolution magnetization prepared rapid acquisition gradient echo (MPRAGE) images with 1 x 1 x 1 mm3 isotropic voxels. For the stimuli-exposed image acquisitions, T2*-weighted gradient-echo echo-planar imaging (GE-EPI) with 1.5 x 1.5 x 2 mm3 voxels will be used. A flip angle of 90 degrees and a bandwidth of 1500 Hz will be used. The field of view will be 192 x 192 mm with a 64 x 64 mm matrix resolution. With this phase encoding, the spatial resolution will be 3 mm, with an echo time (TE) of 25 ms, a repetition time (TR) of 2.5 s, and a multi-slice imaging factor of 2 being employed. With these parameters, 170 volumes will be captured. To un-distort images, the GE-EPI fMRI data will be mapped to a non-distorted set of GE images from the same participant. Next, the non-distorted GE images will be mapped to the T1-weighted MPRAGE image. Finally, the T1-weighted MPRAGE will be mapped to the Montreal Neurological Institute (MNI) standardized brain template. In doing this, the GE-EPI fMRI data will be mapped to the MNI template with maximum accuracy.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 diagnosis of OCD made by a psychiatrist on the research team
* Competence to consent to participate
* Ability to speak and read English
* Consistent and reliable access to the internet

Exclusion Criteria:

* Metal implants
* Active psychosis
* Acute mania
* Severe alcohol or substance use disorder
* Active suicidal or homicidal ideation
* Receiving any additional form of psychotherapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-07-28 (Actual)

PRIMARY OUTCOMES:
Changes in Brain Structure and Activation: Functional Magnetic Resonance Imaging (fMRI) | Week 1, Week 16
  fMRI will be administered to observe any changes in structure.
Changes in symptoms: Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) | Week 1, Week 8, Week 16, 6 Months
  Y-BOCS will be administered to analyze changes in symptoms from treatment. Scale of 0-4 for each question with 0 being no symptom severity and 4 being high symptom severity
Changes in symptoms: Obsessive-Compulsive Inventory - Revised (OCI-R) | Week 1, Week 8, Week 16, 6 months
  OCI-R will be administered to analyze changes in symptoms from treatment. Scale of 0-4 with 0 being not at all and 4 being extreme severity.
Changes in Quality of Life: Quality of Life and Enjoyment Questionnaire (Q-LES-Q) | Week 1, Week 8, Week 16, 6 months
  Q-LES-Q will be administered to analyze changes in quality of life from treatment. Scale of 0-5 for each question with 0 being not at all and 5 being frequently
Changes in level of functioning: Sheehan Disability Scale (SDS0 | Week 1, Week 8, Week 16, 6 Months
  SDS will be administered to analyze changes in levels of functioning. Scale of 0-10, 10 being the worst.

CONTACTS AND LOCATIONS:
Overall Officials: Callum Stephenson, BScH, Principal Investigator — Queen's University
Locations (1):
- Queen's University, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Only care providers involved in care of participants will have access to their information. Participants will only be identifiable by an ID number on the OPTT platform. Only anonymized data will be provided to the analysis team members. All data is encrypted by OPTT and no employee has direct access to patient data.

REFERENCES:
- [Derived] Stephenson C, Malakouti N, Nashed JY, Salomons T, Cook DJ, Milev R, Alavi N. Using Electronically Delivered Therapy and Brain Imaging to Understand Obsessive-Compulsive Disorder Pathophysiology: Protocol for a Pilot Study. JMIR Res Protoc. 2021 Sep 14;10(9):e30726. doi: 10.2196/30726. PMID 34348889